CLINICAL TRIAL: NCT01292447
Title: A Randomized Controlled Trial of 2% Lidocaine Gel for IUD Insertion
Brief Title: A Trial of 2% Lidocaine Gel for Intrauterine Device (IUD) Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Rebecca H. Allen, MD, Assistant Professor ob/gyn, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10-0084
Record Dates: First submitted 2011-01-24; First posted 2011-02-09 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Pain
Keywords: Pain measurement; Intrauterine devices; Lidocaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Will receive placement of inert glycerin gel on ectocervix and in cervical canal prior to IUD placement.
  Interventions: Drug: Placebo gel
- Study Group (Experimental): Will receive placement of 2% lidocaine gel on ectocervix and in cervical canal prior to IUD placement.
  Interventions: Drug: 2% lidocaine gel

INTERVENTIONS:
Drug: 2% lidocaine gel — 120mg lidocaine x 1
  Arms: Study Group
Drug: Placebo gel — Inert gel x 1
  Arms: Control Group

SUMMARY:
The intrauterine device (IUD) is a long-acting, highly effective, reversible contraceptive that may be underutilized due to fear of pain during insertion. Although providers frequently prescribe non-steroidal anti-inflammatory drugs (NSAIDs) for IUD insertion, there is no evidence for any pain reduction. In fact, no interventions evaluated in randomized controlled trials have been shown to be effective in reducing pain during IUD insertion. While many women tolerate IUD insertion well, others have moderate to severe pain. This double-blind randomized controlled trial of 150 women aims to estimate the efficacy of intracervical 2% lidocaine gel compared to placebo (KY jelly) to reduce IUD insertion pain. Our hypothesis is that women who are treated with 2% lidocaine gel prior to IUD insertion will have reduced pain as measured on a 0 mm to 100 mm Visual Analog Scale (VAS). We will be able to detect a 15 mm difference on the VAS with our sample size. Other data to be collected include information regarding age, BMI, obstetric history, lactation status, time since pregnancy or delivery, last menstrual period, history of cervical conization, anxiety levels, anticipated pain levels, insertion characteristics (time, difficulty, complications), side effects, and satisfaction with pain control. If 2% lidocaine gel is effective, then a viable, easily administered option for pain control will be available to providers and patients.

ELIGIBILITY:
Inclusion Criteria:

1. plans for IUD insertion for contraception or abnormal uterine bleeding;
2. 18 to 49 years of age;
3. reached more than 6 weeks postpartum or 2 weeks postabortion if recently pregnant;
4. no prior IUD use;
5. not taken analgesics or anxiolytics in the previous 24 hours;
6. not taken misoprostol prior to IUD insertion;
7. the ability and are willing to give informed consent;
8. speaks English or Spanish.

Exclusion Criteria:

1. any contraindication to IUD placement;
2. allergy to lidocaine or sensitivities to components of the lidocaine or placebo gel;
3. chronic narcotic/benzodiazepine/barbiturate use within the past year.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca H Allen, MD, MPH, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (2):
- United States (2):
  - Women's Primary Care Center/Women and Infants' Hospital, Providence, Rhode Island
  - Womens Primary Care Center, Providence, Rhode Island

REFERENCES:
- [Derived] Allen RH, Raker C, Goyal V. Higher dose cervical 2% lidocaine gel for IUD insertion: a randomized controlled trial. Contraception. 2013 Dec;88(6):730-6. doi: 10.1016/j.contraception.2013.07.009. Epub 2013 Aug 1. PMID 24012096

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 75 | 75
Completed | 73 | 72
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5) | 26.2 (5.3) | 25.7 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 72 | 145
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score During IUD Insertion
Description: 0 to 100 mm visual analog scale, higher values represent more pain.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 73 | 72
score on a scale | 36.7 (30) | 35.2 (27.7)

ADVERSE EVENTS:
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 1/73 | 1/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=73) | Study Group (N=72)
Acute complication (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes